CLINICAL TRIAL: NCT05259189
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of NBL-012 in Healthy Chinese Subjects
Brief Title: A Study of NBL-012 in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NovaRock Biotherapeutics, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: NBL-012-CSP-001
Record Dates: First submitted 2022-01-29; First posted 2022-02-28 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NBL-012 Injection (Experimental): Two subjects will be enrolled in the initial dose. 8 out of 10 healthy subjects will be randomized to receive a single dose of NBL-012 Injection for subsequent dose cohorts
  Interventions: Drug: NBL-012 Injection
- Placebo (Placebo Comparator): 2 out of 10 healthy subjects will be randomized to receive a single dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NBL-012 Injection — a single subcutaneous injection
  Arms: NBL-012 Injection
Drug: Placebo — a single subcutaneous injection
  Arms: Placebo

SUMMARY:
This is a phase 1, randomized, double-blind, placebo-controlled, sequential cohort study to evaluate the safety, tolerability and pharmacokinetics (PK) of NBL-012 as single ascending doses (SAD) administered subcutaneously to healthy Chinese subjects.

DETAILED DESCRIPTION:
This is a phase 1, randomized, double-blind, placebo-controlled, sequential cohort study to evaluate the safety, tolerability and pharmacokinetics of NBL-012 administered subcutaneously as single ascending doses (SAD) to healthy Chinese subjects. Six dose cohorts will be intended for enrollment. The first dose will be sentinel group which will consist of 2 subjects, both of whom will receive active NBL-012. For subsequent dose cohorts, subjects will be given a single escalating SC dose of NBL-01

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and/or female subjects between the ages of 18 and 45 years (inclusive) at screening.
2. Body Mass Index (BMI) of 18 to 26 kg/m2 (inclusive), body weight for male ≥50 kg and for female≥45 kg.
3. Good general health defined as no clinically significant abnormalities identified by a detailed medical history (thoracic and abdominal examination, nervous and mental system examination, etc.), full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG,

Exclusion Criteria:

1. Participated in any drug or medical device clinical trial within 3 months before screening
2. Pregnant or nursing (lactating) women who have a positive blood/urine pregnancy test.
3. Females of child-bearing potential (defined as all females physiologically capable of becoming pregnant) and males who are unwilling or unable to use effective contraception during the study and until the end of study visit (more than 15 weeks after drug administration), or subjects with a plan to give birth wi

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Up to Day 113 from screening
  Number of participants with treatment-related adverse events will be assessed by CTCAE v5.0. The AEs will be summarized according to the system organ class (SOC) and preferred term (PT), including the number and percentage of participants who had AEs.
Clinically significant changes from baseline in 12-lead electrocardiogram (ECG) examination will be recorded as AEs at each visit time point. | Up to Day 113 from screening
  ECG monitoring includes heart rate in bpm.
Clinically significant changes from baseline in 12-lead electrocardiogram (ECG) examination will be recorded as AEs at each visit time point. | Up to Day 113 from screening
  ECG monitoring includes P-R, QT and QTc intervals in ms.
Clinically significant changes from baseline in physical examination will be recorded as AEs at each visit time point. | Up to Day 113 from screening
  Physical examination includes general conditions, skin, neck, chest, spine, limbs, nervous system, and lymphatic system.
Clinically significant changes from baseline in vital signs examination will be recorded as AEs at each visit time point. | Up to Day 113 from screening
  Vital signs monitoring includes body temperature in degrees Celsius.
Clinically significant changes from baseline in vital signs examination will be recorded as AEs at each visit time point. | Up to Day 113 from screening
  Vital signs monitoring includes respiratory rate and pulse in times per minute.
Clinically significant changes from baseline in vital signs examination will be recorded as AEs at each visit time point. | Up to Day 113 from screening
  Vital signs monitoring includes systolic blood pressure and diastolic blood pressure in mmHg.
Clinically significant changes from baseline in routine blood test will be recorded as AEs at each visit time point. | Up to Day 113 from screening
  Routine blood test includes white blood cell count, platelet, neutrophilic granulocyte count, lymphocyte count and monocyte count in 10^9 /L.
Clinically significant changes from baseline in blood biochemistry test will be recorded as AEs at each visit time point. | Up to Day 113 from screening
  Blood biochemistry test includes alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase and glutamyltranspeptidase in U/L.
Clinically significant changes from baseline in routine urine test will be recorded as AEs at each visit time point. | Up to Day 113 from screening
  Routine urine test includes glucose and protein in mg/dL.

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) of NBL-012 injection | Pre-dose and multiple timepoints up to 113 days post-dose
Area under the plasma concentration versus time curve (AUC) of NBL-012 injection | Pre-dose and multiple timepoints up to 113 days post-dose
Time to achieve maximum plasma concentration (Tmax) of NBL-012 injection | Pre-dose and multiple timepoints up to 113 days post-dose
Apparent clearance(CL/F) of NBL-012 injection | Pre-dose and multiple timepoints up to 113 days post-dose
Apparent volume of Distribution(Vz/F) of NBL-012 injection | Pre-dose and multiple timepoints up to 113 days post-dose
Half-life(t1/2) of NBL-012 injection | Pre-dose and multiple timepoints up to 113 days post-dose
The incidence of Anti-drug antibody (ADA) | Pre-dose and multiple timepoints up to 113 days post-dose
  The incidence of Anti-drug antibody (ADA)
Free IL-23 concentration in Serum. | Pre-dose and multiple timepoints up to 113 days post-dose
  Free IL-23 concentration in Serum.

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miu, MD PhD, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University., Suzhou, Jiangsu, China